CLINICAL TRIAL: NCT07214727
Title: A Phase 1, Randomized, Placebo-controlled Study With a Double Blind Period With Open-label Extension Period to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intrathecally Administered ALN-5288 in Adult Patients With Alzheimer's Disease
Brief Title: A Study to Evaluate ALN-5288 in Patients With Alzheimer's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALN-5288-001; 2025-522582-30-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Alzheimer's Disease
Keywords: AD; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ALN-5288 (Experimental): Participants will be administered ALN-5288 in the Double-blind (DB) Period and Open-Label Extension (OLE) Period.
  Interventions: Drug: ALN-5288
- Placebo + ALN-5288 (Placebo Comparator): Participants will be administered placebo in the DB Period and ALN-5288 in the OLE Period.
  Interventions: Drug: ALN-5288; Drug: Placebo

INTERVENTIONS:
Drug: ALN-5288 — ALN-5288 will be administered IT.
Drug: Placebo — Placebo will be administered IT.
  Arms: Placebo + ALN-5288

SUMMARY:
The purpose of this study is to:

* Evaluate the safety and tolerability of intrathecal (IT) ALN-5288 in patients with Alzheimer's Disease (AD)
* Evaluate the pharmacodynamic (PD) and pharmacokinetic (PK) effects of ALN-5288 after dose administration

ELIGIBILITY:
Inclusion Criteria:

* Is able and willing to meet all study requirements in the opinion of the Investigator
* Has a diagnosis of Alzheimer's disease (AD) based on clinical findings supported by cerebrospinal fluid (CSF) biomarkers or positive positron emission tomography (PET) amyloid imaging within 7 years prior to screening
* Has mild cognitive impairment (MCI) or dementia due to AD

Exclusion Criteria:

* Has non-AD dementia
* Has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >2× upper limit of normal (ULN)
* Has total bilirubin >1.5×ULN
* Has known human immunodeficiency virus infection
* Has history of hepatitis C virus or current hepatitis B virus infection
* Has systolic blood pressure >160 mmHg and/or a diastolic blood pressure >100 mmHg after 10 minutes of rest at screening
* Has an estimated glomerular filtration (eGFR) of <45 mL/min/1.73 m^2 at screening
* Has clinically significant ECG abnormalities at screening
* Has uncontrolled psychiatric disease, including patients deemed by the Investigator to be at significant risk of suicide, major depressive episode, psychosis, confusional state, or violent behavior
* Has history of bleeding diathesis or coagulopathy due to chronic conditions
* Has a medical history of brain or spinal disease that would interfere with the IT injection and LP procedures
* Has history of uncontrolled seizures within the last 6 months prior to Screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) | Up to 32 months
Severity of AEs | Up to 32 months

SECONDARY OUTCOMES:
Concentration of Total Tau (t-Tau) Protein in CSF Over Time | Up to 32 months
Change from Baseline in Concentration of t-Tau Protein in CSF Over Time | Up to 32 months
Concentration of ALN-5288 in Plasma Over Time (Ct) | Up to 32 months
Change from Baseline in Concentration of ALN-5288 CSF Ct | Up to 32 months
Concentration of ALN-5288 in Plasma | Up to 32 months
Concentration of ALN-5288 in Urine | Up to 32 months
Concentration of ALN-5288 in CSF | Up to 32 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals Inc
Locations (12):
- Canada (3):
  - Clinical Trial Site, Ottawa, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Montreal, Quebec
- Clinical Trial Site, Amsterdam, Netherlands
- Spain (3):
  - Clinical Trial Site, Barcelona, B
  - Clinical Trial Site, Sant Cugat del Vallès, B
  - Clinical Trial Site, Madrid
- United Kingdom (5):
  - Clinical Trial Site, Southampton, HAM
  - Clinical Trial Site, London, LND
  - Clinical Trial Site, Glasgow
  - Clinical Trial Site, Manchester
  - Clinical Trial Site, Sheffield

IPD SHARING:
Plan to Share IPD: No